CLINICAL TRIAL: NCT03775564
Title: Effectiveness of the RemedRugby Program, a Program of Ecological Cognitive Remediation of Social Cognition Disorders in Schizophrenia
Brief Title: Effectiveness of the RemedRugby Program
Acronym: RemedRugby
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Center Alpes-Isère (Other)
Collaborators: Centre Hospitalier Le Valmont (Valence) (Unknown); Hôpital le Vinatier (Other); Centre Hospitalier Spécialisé de la Savoie (Chambéry) (Unknown); Centre Hospitalier Annecy Genevois (Other); Centre Hospitalier Universitaire de Saint Etienne (Other); Centre Hospitalier Sainte Marie de Clermont Ferrand (Unknown); University Hospital, Clermont-Ferrand (Other)
Responsible Party: Principal Investigator, Dr Julien Dubreucq, Medical Doctor, Hospital Center Alpes-Isère
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-A01612-45
Record Dates: First submitted 2018-07-27; First posted 2018-12-14 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Schizophrenia; Social Cognition; Self Esteem; Empowerment; Recovery
MeSH Terms: conditions — Schizophrenia; Empowerment

STUDY DESIGN:
Intervention Model Description: RemedRugby program Vs TAU + TouchRugby
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REMEDRUGBY (Experimental): TAU + RemedRugby Program
  Interventions: Other: REMEDRUGBY PROGRAM; Other: TAU
- TAU + TOUCH RUGBY (Active Comparator): TAU + Touch Rugby Program
  Interventions: Other: TOUCH RUGBY PROGRAM; Other: TAU

INTERVENTIONS:
Other: REMEDRUGBY PROGRAM — * 1st Session presentation of the programme, its objectives and a common reflection on the concepts of stigmatization/destigmatization.
  * 2nd to 4th session devoted to a group reflection on social conventions and their meaning followed by a practice by means of role-playing.
  * 5th to 7th session devoted to writing comments about tournaments on the blog by working on the intentions of others and the emotional impact of comments on their recipients.
  * 8th, 9th 11th sessions devoted to media relations with group reflection on the image of themselves and their pathology that participants wish to refer to the media, followed by a practice in role-playing games Interviewer-interviewed
  * 10th session devoted to planning and organizing the day of matches with writing a program of the day and spreading on the blog
  * 12th General Debriefing session Including : - 3 tournaments
  * 8 hours of Touch Rugby
  Arms: REMEDRUGBY
Other: TOUCH RUGBY PROGRAM — Practical training Program at Touchrugby at the rate of 12 weekly sessions of 2 hours and 3 inter-institutional tournaments per day
  Arms: TAU + TOUCH RUGBY
Other: TAU — Treatment as usual

SUMMARY:
REMEDRUGBY's objective is to strengthen the capacity of users to interact with others in an assertive way and to fight against stigma. It proposes to specifically target the processes of "social cognition".

"Social cognition" brings together the mental mechanisms that allow everyone to decipher the social situations, emotions and intentions of others and interact with others in the different contexts of everyday life.

People with a psychic handicap frequently have difficulties in this area, which has often important consequences for their social and professional integration.

The REMEDRUGBY program proposes to work specifically on these processes in the context of sport (+ role Play and blog) to strengthen the ability to interact with others and to deal with the stigma that can be encountered on a daily basis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia, schizo-affective disorder (DSM-V criteria; APA, 2013).
* French mother tongue.
* psychotropic treatment unchanged during the month prior to inclusion.
* Patients who gave their informed consent to participate in the study.
* affiliated with a social security scheme or beneficiary of such a scheme
* Subject suitable for the practice of sport.

Exclusion Criteria:

* Recent dependence and abuse on cannabis or any other substance (DSM-V criteria), except tobacco.
* Neurological disorders of vascular, infectious or neurodegenerative origin.
* taking of medicinal products with a cerebral or psychic impact (e.g., corticosteroids).
* Inability to practice sport
* Pregnancy planned or in progress
* Simultaneous Participation in any other program of remediation of social cognition, training in social skills, self-esteem.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Movie to Assess Social Cognition (MASC) | Changes between baseline function, after intervention and at 6 months of follow-up
  Changes in the aggregates (average) of standardized performance levels : z-scores of Theory of Mind (range 0-45) during social cognitive remediation

SECONDARY OUTCOMES:
Positive and Negative Symptoms Scale for Schizophrenia (PANSS) | Changes between baseline function, after intervention and at 6 months of follow-up
  Changes in the aggregates (average) of standardized performance levels : z-scores of positive and negative symptoms (minimum score 30- maximum score 210) of schizophrenia after social cognitive remediation
Personal and Social Performance scale (PSP) | Changes between baseline function, after intervention and at 6 months of follow-up
  Changes in the aggregates (average) of standardized performance levels : z-scores of social function (0 to 100) after social cognitive remediation
Self Esteem Rating Scale (SERS) | Changes between baseline function, after intervention and at 6 months of follow-up
  Changes in the aggregates (average) of standardized performance levels : z-scores (minimum score 10-maximum score 70) in self-assessment of self-esteem
Boston University Empowerment Scale (BUES) | Changes between baseline function, after intervention and at 6 months of follow-up
  Changes in the aggregates (average) of standardized performance levels : z-scores (minimum score 1- maximum score 4) in self-assessment of empowerment
Internalized Stigma of Mental Illness (ISMI) | Changes between baseline function, after intervention and at 6 months of follow-up
  self-assessment of internalized stigma
Stages of Recovery Instrument (STORI) | Changes between baseline function, after intervention and at 6 months of follow-up
  Self-assessment of personal recovery
Social Perception and Knowledge (PerSo) | Changes between baseline function, after intervention and at 6 months of follow-up
  cognitive task to assess competence in perception of social situations and social knowledge
Ambiguous Intentions and Hostility Questionnaire (AIHQ) | Changes between baseline function, after intervention and at 6 months of follow-up
  Changes in the aggregates (average) of standardized performance levels : z-scores (minimum score 1, maximum score 6) at a cognitive task to measure hostile social cognitive bias
Questionnaire of Cognitive and Affective Empathy | Changes between baseline function, after intervention and at 6 months of follow-up
  Changes in the aggregates (average) of standardized performance levels : z-scores (minimum score 31, maximum score 124) in a self-assessment of empathy
French National Adult Reading Test (f-NART | Baseline measure only
  cognitive task to assess premorbid intellectual quotient (IQ)
Trail Making Test A (TMT A) | Changes between baseline function, after intervention and at 6 months of follow-up
  cognitive task to assess speed of processing
Trail Making Test B (TMT B) | Changes between baseline function, after intervention and at 6 months of follow-up
  cognitive task to assess reactive mental flexibility
Self-assessment of Social Cognition (AcSo) | Changes between baseline function, after intervention and at 6 months of follow-up
  self-assessment of patient' perception of social cognitive deficits
Commission Test (modified zoo test) | Changes between baseline function, after intervention and at 6 months of follow-up
  cognitive task to asess planification abilities

CONTACTS AND LOCATIONS:
Overall Officials: Julien JD DUBREUCQ, MD, Principal Investigator — Hospital Center Alpes-Isère
Locations (8):
- France (8):
  - Ch Annecy-Genevois, Annecy, AURA
  - Ch Le Vinatier, Bron, Aura
  - Chs de La Savoie, Chambéry, AURA
  - Ch Sainte-Marie, Clermont-Ferrand, AURA
  - CHU de CLERMONT-FERRAND, Clermont-Ferrand, AURA
  - Chu Saint-Etienne, Saint-Etienne, AURA
  - HCAlpesIsere, Saint-Égrève, AURA
  - Chs Le Valmont, Valence, AURA

REFERENCES:
- [Background] Abu-Akel A. A neurobiological mapping of theory of mind. Brain Res Brain Res Rev. 2003 Sep;43(1):29-40. doi: 10.1016/s0165-0173(03)00190-5. PMID 14499460
- [Background] Addington J, Addington D. Neurocognitive and social functioning in schizophrenia: a 2.5 year follow-up study. Schizophr Res. 2000 Jul 7;44(1):47-56. doi: 10.1016/s0920-9964(99)00160-7. PMID 10867311
- [Background] Addington J, Saeedi H, Addington D. Influence of social perception and social knowledge on cognitive and social functioning in early psychosis. Br J Psychiatry. 2006 Oct;189:373-8. doi: 10.1192/bjp.bp.105.021022. PMID 17012662
- [Background] Aleman A, Hijman R, de Haan EH, Kahn RS. Memory impairment in schizophrenia: a meta-analysis. Am J Psychiatry. 1999 Sep;156(9):1358-66. doi: 10.1176/ajp.156.9.1358. PMID 10484945
- [Background] Baudouin JY, Martin F, Tiberghien G, Verlut I, Franck N. Selective attention to facial emotion and identity in schizophrenia. Neuropsychologia. 2002;40(5):503-11. doi: 10.1016/s0028-3932(01)00114-2. PMID 11749980
- [Background] Baron-Cohen S, Leslie AM, Frith U. Does the autistic child have a "theory of mind"? Cognition. 1985 Oct;21(1):37-46. doi: 10.1016/0010-0277(85)90022-8. No abstract available. PMID 2934210
- [Background] Bellack AS, Brown SA. Psychosocial treatments for schizophrenia. Curr Psychiatry Rep. 2001 Oct;3(5):407-12. doi: 10.1007/s11920-996-0035-x. PMID 11559478
- [Background] Bentall RP, Corcoran R, Howard R, Blackwood N, Kinderman P. Persecutory delusions: a review and theoretical integration. Clin Psychol Rev. 2001 Nov;21(8):1143-92. doi: 10.1016/s0272-7358(01)00106-4. PMID 11702511
- [Background] Bengtsson-Tops A. Mastery in patients with schizophrenia living in the community: relationship to sociodemographic and clinical characteristics, needs for care and support, and social network. J Psychiatr Ment Health Nurs. 2004 Jun;11(3):298-304. doi: 10.1111/j.1365-2850.2003.00718.x. PMID 15149377
- [Background] Bertrand MC, Sutton H, Achim AM, Malla AK, Lepage M. Social cognitive impairments in first episode psychosis. Schizophr Res. 2007 Sep;95(1-3):124-33. doi: 10.1016/j.schres.2007.05.033. Epub 2007 Jul 16. PMID 17630261
- [Background] Blair RJ. Responding to the emotions of others: dissociating forms of empathy through the study of typical and psychiatric populations. Conscious Cogn. 2005 Dec;14(4):698-718. doi: 10.1016/j.concog.2005.06.004. Epub 2005 Sep 12. PMID 16157488
- [Background] Blanchard JJ, Mueser KT, Bellack AS. Anhedonia, positive and negative affect, and social functioning in schizophrenia. Schizophr Bull. 1998;24(3):413-24. doi: 10.1093/oxfordjournals.schbul.a033336. PMID 9718633
- [Background] Bora E, Yucel M, Pantelis C. Theory of mind impairment in schizophrenia: meta-analysis. Schizophr Res. 2009 Apr;109(1-3):1-9. doi: 10.1016/j.schres.2008.12.020. Epub 2009 Feb 4. PMID 19195844
- [Background] Ritsher JB, Otilingam PG, Grajales M. Internalized stigma of mental illness: psychometric properties of a new measure. Psychiatry Res. 2003 Nov 1;121(1):31-49. doi: 10.1016/j.psychres.2003.08.008. PMID 14572622
- [Background] Brohan E, Elgie R, Sartorius N, Thornicroft G; GAMIAN-Europe Study Group. Self-stigma, empowerment and perceived discrimination among people with schizophrenia in 14 European countries: the GAMIAN-Europe study. Schizophr Res. 2010 Sep;122(1-3):232-8. doi: 10.1016/j.schres.2010.02.1065. Epub 2010 Mar 26. PMID 20347271
- [Background] Brune M. "Theory of mind" in schizophrenia: a review of the literature. Schizophr Bull. 2005 Jan;31(1):21-42. doi: 10.1093/schbul/sbi002. Epub 2005 Feb 16. PMID 15888423
- [Background] Chang WC, Hui CL, Tang JY, Wong GH, Lam MM, Chan SK, Chen EY. Persistent negative symptoms in first-episode schizophrenia: a prospective three-year follow-up study. Schizophr Res. 2011 Dec;133(1-3):22-8. doi: 10.1016/j.schres.2011.09.006. Epub 2011 Oct 2. PMID 21968080
- [Background] Choi J, Fiszdon JM, Medalia A. Expectancy-value theory in persistence of learning effects in schizophrenia: role of task value and perceived competency. Schizophr Bull. 2010 Sep;36(5):957-65. doi: 10.1093/schbul/sbq078. Epub 2010 Jul 15. PMID 20634277
- [Background] Combs DR, Adams SD, Penn DL, Roberts D, Tiegreen J, Stem P. Social Cognition and Interaction Training (SCIT) for inpatients with schizophrenia spectrum disorders: preliminary findings. Schizophr Res. 2007 Mar;91(1-3):112-6. doi: 10.1016/j.schres.2006.12.010. Epub 2007 Feb 12. PMID 17293083
- [Background] Corcoran R, Mercer G, Frith CD. Schizophrenia, symptomatology and social inference: investigating "theory of mind" in people with schizophrenia. Schizophr Res. 1995 Sep;17(1):5-13. doi: 10.1016/0920-9964(95)00024-g. PMID 8541250
- [Background] Corcoran R, Rowse G, Moore R, Blackwood N, Kinderman P, Howard R, Cummins S, Bentall RP. A transdiagnostic investigation of 'theory of mind' and 'jumping to conclusions' in patients with persecutory delusions. Psychol Med. 2008 Nov;38(11):1577-83. doi: 10.1017/S0033291707002152. Epub 2007 Nov 16. PMID 18005499
- [Background] Couture SM, Penn DL, Roberts DL. The functional significance of social cognition in schizophrenia: a review. Schizophr Bull. 2006 Oct;32 Suppl 1(Suppl 1):S44-63. doi: 10.1093/schbul/sbl029. Epub 2006 Aug 17. PMID 16916889
- [Background] Couture SM, Granholm EL, Fish SC. A path model investigation of neurocognition, theory of mind, social competence, negative symptoms and real-world functioning in schizophrenia. Schizophr Res. 2011 Feb;125(2-3):152-60. doi: 10.1016/j.schres.2010.09.020. Epub 2010 Oct 20. PMID 20965699
- [Background] Darba J, Minoves A, Rojo E, Jimenez F, Rejas J. Efficacy of second-generation-antipsychotics in the treatment of negative symptoms of schizophrenia: a meta-analysis of randomized clinical trials. Rev Psiquiatr Salud Ment. 2011 Jul;4(3):126-43. doi: 10.1016/j.rpsm.2011.02.005. Epub 2011 Jun 14. English, Spanish. PMID 23446193
- [Background] de Haan L, Linszen DH, Lenior ME, de Win ED, Gorsira R. Duration of untreated psychosis and outcome of schizophrenia: delay in intensive psychosocial treatment versus delay in treatment with antipsychotic medication. Schizophr Bull. 2003;29(2):341-8. doi: 10.1093/oxfordjournals.schbul.a007009. PMID 14552508
- [Background] Demily C, Franck N. Cognitive remediation: a promising tool for the treatment of schizophrenia. Expert Rev Neurother. 2008 Jul;8(7):1029-36. doi: 10.1586/14737175.8.7.1029. PMID 18590474
- [Background] Deutsch F, Madle RA. Empathy: historic and current conceptualizations, measurement, and a cognitive theoretical perspective. Hum Dev. 1975;18(4):267-87. doi: 10.1159/000271488. No abstract available. PMID 765261
- [Background] Dziobek I, Rogers K, Fleck S, Bahnemann M, Heekeren HR, Wolf OT, Convit A. Dissociation of cognitive and emotional empathy in adults with Asperger syndrome using the Multifaceted Empathy Test (MET). J Autism Dev Disord. 2008 Mar;38(3):464-73. doi: 10.1007/s10803-007-0486-x. Epub 2007 Nov 8. PMID 17990089
- [Background] Edwards J, Jackson HJ, Pattison PE. Emotion recognition via facial expression and affective prosody in schizophrenia: a methodological review. Clin Psychol Rev. 2002 Jul;22(6):789-832. doi: 10.1016/s0272-7358(02)00130-7. PMID 12214327
- [Background] Fett AK, Viechtbauer W, Dominguez MD, Penn DL, van Os J, Krabbendam L. The relationship between neurocognition and social cognition with functional outcomes in schizophrenia: a meta-analysis. Neurosci Biobehav Rev. 2011 Jan;35(3):573-88. doi: 10.1016/j.neubiorev.2010.07.001. Epub 2010 Jul 8. PMID 20620163
- [Background] Jolley S, Garety P, Bebbington P, Dunn G, Freeman D, Kuipers E, Fowler D, Hemsley D. Attributional style in psychosis--the role of affect and belief type. Behav Res Ther. 2006 Nov;44(11):1597-607. doi: 10.1016/j.brat.2005.12.002. Epub 2006 Jan 24. PMID 16436270
- [Background] Frith CD. Schizophrenia and theory of mind. Psychol Med. 2004 Apr;34(3):385-9. doi: 10.1017/s0033291703001326. No abstract available. PMID 15259823
- [Background] Galderisi S, Bucci P, Mucci A, Kirkpatrick B, Pini S, Rossi A, Vita A, Maj M. Categorical and dimensional approaches to negative symptoms of schizophrenia: focus on long-term stability and functional outcome. Schizophr Res. 2013 Jun;147(1):157-162. doi: 10.1016/j.schres.2013.03.020. Epub 2013 Apr 19. PMID 23608244
- [Background] Galderisi S, Mucci A, Bitter I, Libiger J, Bucci P, Fleischhacker WW, Kahn RS; Eufest Study Group. Persistent negative symptoms in first episode patients with schizophrenia: results from the European First Episode Schizophrenia Trial. Eur Neuropsychopharmacol. 2013 Mar;23(3):196-204. doi: 10.1016/j.euroneuro.2012.04.019. Epub 2012 May 28. PMID 22647933
- [Background] Green MF, Olivier B, Crawley JN, Penn DL, Silverstein S. Social cognition in schizophrenia: recommendations from the measurement and treatment research to improve cognition in schizophrenia new approaches conference. Schizophr Bull. 2005 Oct;31(4):882-7. doi: 10.1093/schbul/sbi049. Epub 2005 Aug 31. PMID 16135561
- [Background] Green MF, Penn DL, Bentall R, Carpenter WT, Gaebel W, Gur RC, Kring AM, Park S, Silverstein SM, Heinssen R. Social cognition in schizophrenia: an NIMH workshop on definitions, assessment, and research opportunities. Schizophr Bull. 2008 Nov;34(6):1211-20. doi: 10.1093/schbul/sbm145. Epub 2008 Jan 8. PMID 18184635
- [Background] Green MF, Leitman DI. Social cognition in schizophrenia. Schizophr Bull. 2008 Jul;34(4):670-2. doi: 10.1093/schbul/sbn045. Epub 2008 May 20. PMID 18495642
- [Background] Hardy-Bayle MC, Sarfati Y, Passerieux C. The cognitive basis of disorganization symptomatology in schizophrenia and its clinical correlates: toward a pathogenetic approach to disorganization. Schizophr Bull. 2003;29(3):459-71. doi: 10.1093/oxfordjournals.schbul.a007019. PMID 14609240
- [Background] Kalpakci A, Vanwoerden S, Elhai JD, Sharp C. The Independent Contributions of Emotion Dysregulation and Hypermentalization to the "Double Dissociation" of Affective and Cognitive Empathy in Female Adolescent Inpatients With BPD. J Pers Disord. 2016 Apr;30(2):242-60. doi: 10.1521/pedi_2015_29_192. Epub 2015 Apr 23. PMID 25905730
- [Background] Harrington L, Siegert RJ, McClure J. Theory of mind in schizophrenia: a critical review. Cogn Neuropsychiatry. 2005 Aug;10(4):249-86. doi: 10.1080/13546800444000056. PMID 16571462
- [Background] Harvey PD, Koren D, Reichenberg A, Bowie CR. Negative symptoms and cognitive deficits: what is the nature of their relationship? Schizophr Bull. 2006 Apr;32(2):250-8. doi: 10.1093/schbul/sbj011. Epub 2005 Oct 12. PMID 16221995
- [Background] Hoekert M, Kahn RS, Pijnenborg M, Aleman A. Impaired recognition and expression of emotional prosody in schizophrenia: review and meta-analysis. Schizophr Res. 2007 Nov;96(1-3):135-45. doi: 10.1016/j.schres.2007.07.023. Epub 2007 Sep 4. PMID 17766089
- [Background] Kee KS, Green MF, Mintz J, Brekke JS. Is emotion processing a predictor of functional outcome in schizophrenia? Schizophr Bull. 2003;29(3):487-97. doi: 10.1093/oxfordjournals.schbul.a007021. PMID 14609242
- [Background] Kohler CG, Bilker W, Hagendoorn M, Gur RE, Gur RC. Emotion recognition deficit in schizophrenia: association with symptomatology and cognition. Biol Psychiatry. 2000 Jul 15;48(2):127-36. doi: 10.1016/s0006-3223(00)00847-7. PMID 10903409
- [Background] Jones AP, Happe FG, Gilbert F, Burnett S, Viding E. Feeling, caring, knowing: different types of empathy deficit in boys with psychopathic tendencies and autism spectrum disorder. J Child Psychol Psychiatry. 2010 Nov;51(11):1188-97. doi: 10.1111/j.1469-7610.2010.02280.x. PMID 20633070
- [Background] Lahera G, Benito A, Montes JM, Fernandez-Liria A, Olbert CM, Penn DL. Social cognition and interaction training (SCIT) for outpatients with bipolar disorder. J Affect Disord. 2013 Mar 20;146(1):132-6. doi: 10.1016/j.jad.2012.06.032. Epub 2012 Jul 25. PMID 22840617
- [Background] Lawrence EJ, Shaw P, Baker D, Patel M, Sierra-Siegert M, Medford N, David AS. Empathy and enduring depersonalization: the role of self-related processes. Soc Neurosci. 2007;2(3-4):292-306. doi: 10.1080/17470910701391794. PMID 18633820
- [Background] Lin CH, Huang CL, Chang YC, Chen PW, Lin CY, Tsai GE, Lane HY. Clinical symptoms, mainly negative symptoms, mediate the influence of neurocognition and social cognition on functional outcome of schizophrenia. Schizophr Res. 2013 May;146(1-3):231-7. doi: 10.1016/j.schres.2013.02.009. Epub 2013 Mar 9. PMID 23478155
- [Background] Livingston JD, Boyd JE. Correlates and consequences of internalized stigma for people living with mental illness: a systematic review and meta-analysis. Soc Sci Med. 2010 Dec;71(12):2150-61. doi: 10.1016/j.socscimed.2010.09.030. Epub 2010 Oct 12. PMID 21051128
- [Background] Lysaker PH, Beattie NL, Strasburger AM, Davis LW. Reported history of child sexual abuse in schizophrenia: associations with heightened symptom levels and poorer participation over four months in vocational rehabilitation. J Nerv Ment Dis. 2005 Dec;193(12):790-5. doi: 10.1097/01.nmd.0000188970.11916.76. PMID 16319700
- [Background] MacLeod J, Nelson G. Programs for the promotion of family wellness and the prevention of child maltreatment: a meta-analytic review. Child Abuse Negl. 2000 Sep;24(9):1127-49. doi: 10.1016/s0145-2134(00)00178-2. PMID 11057701
- [Background] Medalia A, Choi J. Cognitive remediation in schizophrenia. Neuropsychol Rev. 2009 Sep;19(3):353-64. doi: 10.1007/s11065-009-9097-y. Epub 2009 May 15. PMID 19444614
- [Background] Medalia A, Saperstein A. The role of motivation for treatment success. Schizophr Bull. 2011 Sep;37 Suppl 2(Suppl 2):S122-8. doi: 10.1093/schbul/sbr063. PMID 21860041
- [Background] Medalia A, Richardson R. What predicts a good response to cognitive remediation interventions? Schizophr Bull. 2005 Oct;31(4):942-53. doi: 10.1093/schbul/sbi045. Epub 2005 Aug 24. PMID 16120830
- [Background] McGuire PK, Shah GM, Murray RM. Increased blood flow in Broca's area during auditory hallucinations in schizophrenia. Lancet. 1993 Sep 18;342(8873):703-6. doi: 10.1016/0140-6736(93)91707-s. PMID 8103821
- [Background] McGurk SR, Twamley EW, Sitzer DI, McHugo GJ, Mueser KT. A meta-analysis of cognitive remediation in schizophrenia. Am J Psychiatry. 2007 Dec;164(12):1791-802. doi: 10.1176/appi.ajp.2007.07060906. PMID 18056233
- [Background] Montag C, Dziobek I, Richter IS, Neuhaus K, Lehmann A, Sylla R, Heekeren HR, Heinz A, Gallinat J. Different aspects of theory of mind in paranoid schizophrenia: evidence from a video-based assessment. Psychiatry Res. 2011 Apr 30;186(2-3):203-9. doi: 10.1016/j.psychres.2010.09.006. Epub 2010 Oct 14. PMID 20947175
- [Background] Nakagami E, Hoe M, Brekke JS. The prospective relationships among intrinsic motivation, neurocognition, and psychosocial functioning in schizophrenia. Schizophr Bull. 2010 Sep;36(5):935-48. doi: 10.1093/schbul/sbq043. Epub 2010 May 12. PMID 20462998
- [Background] Nasrallah H, Morosini P, Gagnon DD. Reliability, validity and ability to detect change of the Personal and Social Performance scale in patients with stable schizophrenia. Psychiatry Res. 2008 Nov 30;161(2):213-24. doi: 10.1016/j.psychres.2007.11.012. Epub 2008 Oct 11. PMID 18848731
- [Background] Penn DL, Spaulding W, Reed D, Sullivan M. The relationship of social cognition to ward behavior in chronic schizophrenia. Schizophr Res. 1996 Jul 5;20(3):327-35. doi: 10.1016/0920-9964(96)00010-2. PMID 8827860
- [Background] Penn DL, Corrigan PW, Bentall RP, Racenstein JM, Newman L. Social cognition in schizophrenia. Psychol Bull. 1997 Jan;121(1):114-32. doi: 10.1037/0033-2909.121.1.114. PMID 9000894
- [Background] Penn D, Roberts DL, Munt ED, Silverstein E, Jones N, Sheitman B. A pilot study of social cognition and interaction training (SCIT) for schizophrenia. Schizophr Res. 2005 Dec 15;80(2-3):357-9. doi: 10.1016/j.schres.2005.07.011. Epub 2005 Aug 31. No abstract available. PMID 16139480
- [Background] Penn DL, Sanna LJ, Roberts DL. Social cognition in schizophrenia: an overview. Schizophr Bull. 2008 May;34(3):408-11. doi: 10.1093/schbul/sbn014. Epub 2008 Mar 28. PMID 18375928